CLINICAL TRIAL: NCT04680975
Title: A Phase 2, Open-label Multicenter Study to Evaluate the Efficacy and Safety of Belumosudil in Subjects With Diffuse Cutaneous Systemic Sclerosis (dcSSc)
Brief Title: Efficacy and Safety of Belumosudil in Subjects With Diffuse Cutaneous Systemic Sclerosis
Acronym: dcSSC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision due to slow enrollment and strategic consideration; not driven by any safety concerns.
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT17634; KD025-215 (Other: Kadmon)
Record Dates: First submitted 2020-12-11; First posted 2020-12-23 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: skin diseases; systemic sclerosis; phase 2; Scleroderma Health Assessment Questionnaire Disability Index; Modified Rodnan Skin Score; Combined Response Index in dcSSc (CRISS); diffuse cutaneous systemic sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Skin Diseases; Scleroderma, Systemic | interventions — belumosudil; KD025

STUDY DESIGN:
Intervention Model Description: Belumosudil 200 mg PO BID
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belumosudil (Experimental): Participants received belumosudil 200 mg tablet orally PO, BID for 52 weeks.
  Interventions: Drug: Belumosudil

INTERVENTIONS:
Drug: Belumosudil — 10 participants with dcSSc received belumosudil 200 mg PO BID for 52 weeks
  Other Names: KD025

SUMMARY:
This was a phase 2, open-label, single-cohort, multicenter trial of belumosudil in participants with Diffuse Cutaneous Systemic Sclerosis (dcSSc). An estimated total of 12 to 15 participants would receive belumosudil 200 milligrams (mg) administered orally (PO) twice daily (BID) for 52 weeks. The primary analysis was at 24 weeks.

DETAILED DESCRIPTION:
The primary objective of this phase 2, open-label, single-cohort, multicenter trial was to evaluate the efficacy of belumosudil 200 mg BID using the Combined Response Index in diffuse cutaneous Systemic Sclerosis (CRISS) after 24 weeks of therapy. The duration of the study was approximately 14 months (4 weeks for screening, 52 weeks of dosing period, and 4 weeks of Follow-up)

Participants who had signed an Institutional Review Board/Independent Ethics Committee-(IRB/IEC)-approved informed consent form (ICF) and met all of the inclusion/exclusion criteria were enrolled. A total of 10 participants at 6 sites received belumosudil 200 mg in tablet form administered PO BID for 52 weeks. The total duration of the study is approximately 14 months: a 4-week screening period, a 52-week treatment period, and a 4-week follow-up.

The primary endpoint was analyzed using Week 24 data.

Efficacy was assessed throughout the 52-week dosing period using:

* Composite Response Index in Systemic Sclerosis (CRISS)
* Modified Rodnan Skin Score (mRSS)
* Pulmonary Function Tests (PFTs)
* Physician Global Assessment
* Patient Global Assessment

Safety was be assessed throughout the study and will include:.

* Physical examinations (PEs)
* Vital sign measurements
* Weight measurements
* Blood sample collection for hematology and chemistry; urinalysis
* Electrocardiograms (ECGs)
* Adverse event (AE) assessments
* Concomitant medication assessments
* Pregnancy testing for females of childbearing potential.

Reasons for discontinuation of treatment because of adverse events were documented. Careful monitoring of all adverse events was carried out. Dosing could be reduced 1 dose level. If the dose was not tolerated, then the participant was discontinued from the study. If there is an interruption of dosing, after 14 days the participant was discontinued from the study.

Participants were given a study drug diary to record the details of each dose of belumosudil 200 mg. Diaries were dispense/collected on each visit. Compliance with dosing was confirmed using participant diaries, which was examined at each visit by site staff to determine if dosing was as instructed per protocol and follow-up.

A 4-Week Safety Follow-up Visit occurred 28 days (± 3 days) after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants greater than or equal to (>=) 18 years old with the diagnosis of dcSSc according to the 2013 American College of Rheumatology and European League Against Rheumatism.
2. Had disease duration (defined as interval from first non Raynaud disease manifestation) of less than or equal to (<=) 6 years.
3. Had mRSS of >=15 but <=40.
4. Had active disease as determined by the Principal Investigator within the 6 months prior to screening.
5. Adequate organ and bone marrow functions evaluated during the 28 days prior to enrollment as follows:

   1. Absolute neutrophil count >= 1.5*10^9/L
   2. Platelet count >= 100*10^9/L
   3. Total bilirubin <= 1.0*upper limit of normal (ULN)
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST), and serum creatinine <= 1.5*ULN.
6. Female participants of childbearing potential had a negative pregnancy test at screening. Females of childbearing potential were defined as sexually mature women without prior hysterectomy or who had any evidence of menses in the past 12 months. However, women who had been amenorrheic for 12 or more months were still considered to be of childbearing potential if the amenorrhea was possibly due to prior chemotherapy, anti-estrogens, or ovarian suppression.

   1. Women of childbearing potential (i.e., menstruating women) must had a negative urine pregnancy test (positive urine tests were to be confirmed by serum test) documented within the 24-hour period prior to the first dose of study drug.
   2. Sexually active women of childbearing potential enrolled in the study agreed to use two forms of accepted methods of contraception during the course of the study and for 3 months after their last dose of study drug. Effective birth control includes (i) intrauterine device plus 1 barrier method; (ii) on stable doses of hormonal contraception for at least 3 months (e.g., oral, injectable, implant, transdermal) plus 1 barrier method; or (iii) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm), or a vasectomized partner.
7. For male participants who were sexually active and who were partners of premenopausal women: agreement to use 2 forms of contraception as in criterion number 6b above during the treatment period and for at least 3 months after the last dose of study drug.
8. Male participants must not donate sperm for 3 months after last dose of study drug.
9. Able to provide written informed consent prior to the performance of any study-specific procedures.

Exclusion Criteria:

1. Participants had corrected QT interval using Fridericia's formula (QTcF) greater than 450 milliseconds.
2. Ongoing use or current use of concomitant medication known to have the potential for QTc prolongation.
3. Female participant who was pregnant or breastfed.
4. Participated in another study with an investigational drug within 28 days of study entry (for studies involving biologics, within 3 half-lives of the biologic).
5. History or other evidence of severe illness or any other conditions that would make the participant, in the opinion of the Investigator, unsuitable for the study.
6. Chronic heart failure with New York Heart Association Classes II, III, or IV.
7. Acute or chronic liver disease (e.g., cirrhosis).
8. Positive human immunodeficiency virus (HIV) test.
9. Active hepatitis C virus (HCV), hepatitis B virus (HBV), or positive whole blood tuberculin test.
10. Diagnosed with any malignancy within 3 years of enrollment, with the exception of basal cell or completely resected squamous cell carcinoma of the skin, resected in situ cervical malignancy, resected breast ductal carcinoma in situ, or low risk prostate cancer after curative resection.
11. Had previous exposure to belumosudil or known allergy/sensitivity to belumosudil, or any other Rho-associated Protein Kinase-2 (ROCK2) inhibitor.
12. Scleroderma renal crisis within 4 months prior to enrollment.
13. Forced vital capacity <= 50% Predicted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California, Los Angeles Medical Center_Site number 104, Los Angeles, California
  - Yale University School of Medicine_Site number 140, New Haven, Connecticut
  - Northwestern University_Site number 124, Chicago, Illinois
  - Columbia University Medical Center_Site number 086, New York, New York
  - University of Utah_Site number 048, Salt Lake City, Utah
  - Virginia Mason Medical Center_Site number 145, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 active sites. A total of 11 participants were screened between 03 Mar 2021 and 23 Nov 2021, of which 1 participant was screen failure due to not meeting eligibility criteria.
Pre-assignment Details: A total of 10 participants were enrolled and treated with belumosudil in the study.
Groups:
- Belumosudil: Participants received belumosudil 200 milligrams (mg) tablet orally (PO), twice a day (BID) for 52 weeks.
Period: Overall Study
Arm/Group | Belumosudil
Started | 10
Completed | 4
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Death | 1
Not completed — Progressive Disease | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on modified intent to treat (mITT) population which included all participants who received at least 1 dose of belumosudil 200 mg.
Groups:
- Belumosudil: Participants received belumosudil 200 mg tablet PO, BID for 52 weeks.
Arm/Group | Belumosudil
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (7.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Combined Response Index in Diffuse Cutaneous Systemic Sclerosis (CRISS) Score at Week 24
Description: CRISS components included the following domains: modified Rodnan skin score (mRSS), forced vital capacity (FVC) percent predicted, physician global assessment, patient global assessment, and scleroderma health assessment questionnaire disability-index (SHAQ-DI). An algorithm determines the predicted probability of improvement from Baseline by incorporating change in the mRSS, FVC percent predicted, physician and patient global assessments, and SHAQ-DI. The outcome is a continuous variable between 0.0 and 1.0 (0 to 100%). A higher score indicated greater probability of improvement. Participants are not considered improved if they develop new onset of renal crisis, new onset or worsening of lung fibrosis, new onset of pulmonary arterial hypertension, new onset of left ventricular failure during the trial. CRISS score greater than 60% is considered the minimally important difference.
Time Frame: Week 24
Population: Analysis was performed on mITT population. Here, overall number of participants analyzed signifies participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belumosudil
Number analyzed (Participants) | 4
score on a scale | 6.65 (12.926)

2. Secondary Outcome: Combined Response Index in Diffuse Cutaneous Systemic Sclerosis (CRISS) Score at Weeks 8, 16, 36, and 52
Description: CRISS components included the following domains: mRSS, FVC percent predicted, physician global assessment, patient global assessment, and SHAQ-DI. An algorithm determines the predicted probability of improvement from Baseline by incorporating change in the mRSS, FVC percent predicted, physician and patient global assessments, and SHAQ-DI. The outcome is a continuous variable between 0.0 and 1.0 (0 to 100%). A higher score indicated greater probability of improvement. Participants are not considered improved if they develop new onset of renal crisis, new onset or worsening of lung fibrosis, new onset of pulmonary arterial hypertension, new onset of left ventricular failure during the trial. CRISS score greater than 60% is considered the minimally important difference.
Time Frame: Week 8, 16, 36 and 52
Population: Analysis was performed on mITT population. Here, "number analyzed" signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belumosudil
Number analyzed (Participants) | 10
score on a scale
  Week 8: number analyzed (Participants) | 7
  Week 8 | 13.97 (24.657)
  Week 16: number analyzed (Participants) | 5
  Week 16 | 20.48 (41.654)
  Week 36: number analyzed (Participants) | 4
  Week 36 | 22.38 (44.715)
  Week 52: number analyzed (Participants) | 4
  Week 52 | 25.49 (49.674)

3. Secondary Outcome: Modified Rodnan Skin Score (mRSS) at Week 24
Description: The mRSS is an accepted clinical measure of the skin thickness. The investigator assessed the thickening of the skin using the modified Rodnan Skin Score through simple palpation on 17 different skin sites in the fingers, hands, forearms, arms, feet, legs, and thighs (bilaterally) and face, chest, and abdomen (singly). Each skin site was rated on a 0 to 3 scale; where 0 = normal skin, 1 = mild thickness, 2 = moderate thickness, and 3 = severe thickness and unable to pinch. Individual skin scores in the 17 body areas were summed and defined as the total mRSS which ranged from 0 (no thickening) to 51 (severe thickening), where higher score indicated more severity of skin thickening/worst outcome.
Time Frame: Week 24
Population: Analysis was performed on mITT population. Here," overall number of participants analyzed" signifies participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belumosudil
Number analyzed (Participants) | 6
score on a scale | 24.2 (11.16)

4. Secondary Outcome: Forced Vital Capacity (FVC) Level at Week 24
Description: FVC was the total amount of air (in liters) exhaled from the lungs during the lung function test measured by spirometer which assessed the change in lung function related to the disease status of an underlying interstitial lung disease.
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Belumosudil
Number analyzed (Participants) | 6
liters | 85.7 (25.28)

5. Secondary Outcome: Physician Global Assessment of Participant's Overall Health Using Visual Analogue Scale (VAS) Score at Week 24
Description: The Physician Global Assessment (reported by the physician) quantified the participant's overall health during the last week based on a VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome.
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belumosudil
Number analyzed (Participants) | 6
score on a scale | 61.2 (30.32)

6. Secondary Outcome: Patient Global Assessment of Participant's Overall Health Using Visual Analogue Scale (VAS) Score at Week 24
Description: The Patient Global Assessment (reported by participant) quantified the participant's overall health during the last week based on a VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome.
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belumosudil
Number analyzed (Participants) | 6
score on a scale | 51.3 (34.54)

7. Secondary Outcome: Scleroderma Health Assessment Questionnaire-Disability Index (SHAQ-DI) Total Score at Week 24
Description: SHAQ-DI included the general health assessment questionnaire-disability index (HAD-DI) assessment and 6 scleroderma-specific VAS items to explore the impact of participant's disease. The general HAD-DI assessment included 8 domains addressing scleroderma related manifestations that contribute to disability. It is a quality of life measure. For each question, level of difficulty was scored from 0 to 3, where 0=no difficulty, 1=some difficulty, 2=much difficulty, 3=unable to do. Some domains in the SHAQ are visual analog scales that are measured first and then changed to a 0-3 scale. SHAQ-DI total score was computed as the sum of domain scores divided by the number of domains answered and it ranged from 0 (no difficulty) to 3 (maximum difficulty), where higher score indicated greater disability/worse functionality.
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belumosudil
Number analyzed (Participants) | 5
score on a scale | 1.750 (1.072)

8. Secondary Outcome: Change From Baseline in Modified Rodnan Skin Thickness Score (mRSS) at Weeks 8, 16, 36, and 52
Description: The mRSS is an accepted clinical measure of the skin thickness. The investigator assessed the thickening of the skin using the modified Rodnan Skin Score through simple palpation on 17 different skin sites in the fingers, hands, forearms, arms, feet, legs, and thighs (bilaterally) and face, chest, and abdomen (singly). Each skin site was rated on a 0 to 3 scale; where 0 = normal skin, 1 = mild thickness, 2 = moderate thickness, and 3 = severe thickness and unable to pinch. Individual skin scores in the 17 body areas were summed and defined as the total mRSS which ranged from 0 (no thickening) to 51 (severe thickening), where higher score indicated more severity of skin thickening/worst outcome. A negative change from baseline demonstrates improvement.
Time Frame: Baseline, Week 8, 16, 36 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belumosudil
Number analyzed (Participants) | 10
score on a scale
  Week 8: number analyzed (Participants) | 9
  Week 8 | -1.2 (2.82)
  Week 16: number analyzed (Participants) | 6
  Week 16 | -1.0 (4.86)
  Week 36: number analyzed (Participants) | 5
  Week 36 | 0.2 (6.57)
  Week 52: number analyzed (Participants) | 4
  Week 52 | -1.0 (8.98)

9. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) Level at Weeks 8, 16, 36, and 52
Description: FVC was the total amount of air (in liters) exhaled from the lungs during the lung function test measured by spirometer which assessed the change in lung function related to the disease status of an underlying interstitial lung disease. Change from Baseline was calculated by subtracting Baseline value from specified values at each reported week (Week 8, 16, 36 and 52).
Time Frame: Baseline, Week 8, 16, 36 and 52
Population: Analysis was performed on the mITT population. Here, "number analyzed" signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Belumosudil
Number analyzed (Participants) | 10
liters
  Week 8: number analyzed (Participants) | 9
  Week 8 | 0.8 (4.15)
  Week 16: number analyzed (Participants) | 7
  Week 16 | 2.9 (4.85)
  Week 36: number analyzed (Participants) | 4
  Week 36 | 3.3 (9.32)
  Week 52: number analyzed (Participants) | 4
  Week 52 | 0.8 (15.52)

10. Secondary Outcome: Change From Baseline in Physician Global Assessment (Reported by the Physician) Quantified of Participant's Overall Health Using Visual Analogue Scale (VAS) Score at Weeks 8, 16, 36, and 52
Description: The Physician Global Assessment (reported by the physician) quantified the participant's overall health during the last week based on a VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome. A positive change from Baseline demonstrated improvement.
Time Frame: Baseline, Week 8, 16, 36 and 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belumosudil
Number analyzed (Participants) | 10
score on a scale
  Week 8: number analyzed (Participants) | 9
  Week 8 | 0.1 (19.04)
  Week 16: number analyzed (Participants) | 6
  Week 16 | 3.5 (19.72)
  Week 36: number analyzed (Participants) | 5
  Week 36 | 7.6 (29.23)
  Week 52: number analyzed (Participants) | 4
  Week 52 | 12.0 (32.22)

11. Secondary Outcome: Change From Baseline in Patient Global Assessment of Participant's Overall Health Using Visual Analogue Scale (VAS) Score at Weeks 8, 16, 36, and 52
Description: The Patient Global Assessment (reported by participant) quantified the participant's overall health during the last week based on a VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome. A positive change from Baseline demonstrated improvement.
Time Frame: Baseline, Week 8, 16, 36 and 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belumosudil
Number analyzed (Participants) | 10
score on a scale
  Week 8: number analyzed (Participants) | 9
  Week 8 | -5.6 (27.68)
  Week 16: number analyzed (Participants) | 6
  Week 16 | -7.2 (17.38)
  Week 36: number analyzed (Participants) | 5
  Week 36 | -3.0 (45.54)
  Week 52: number analyzed (Participants) | 4
  Week 52 | -20.0 (22.82)

12. Secondary Outcome: Change From Baseline in Scleroderma Health Assessment Questionnaire-Disability Index (SHAQ-DI) Total Score at Weeks 8, 16, 36, and 52
Description: SHAQ-DI VAS included the general HAD-DI assessment and 6 scleroderma-specific VAS items to explore the impact of participant's disease. The general HAD-DI assessment included 8 domains addressing scleroderma related manifestations that contribute to disability. It is a quality of life measure. Each activity category consisted of 2 to 3 items. For each question, level of difficulty was scored from 0 to 3, where 0=no difficulty, 1=some difficulty, 2=much difficulty, 3=unable to do. Some domains in the SHAQ are visual analog scales that are measured first and then changed to a 0-3 scale. SHAQ-DI total score was computed as the sum of domain scores divided by the number of domains answered and it ranged from 0 (no difficulty) to 3 (maximum difficulty), where higher score indicated greater disability/worse functionality.
Time Frame: Baseline, Week 8, 16, 36 and 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belumosudil
Number analyzed (Participants) | 10
score on a scale
  Week 8: number analyzed (Participants) | 9
  Week 8 | -0.069 (0.208)
  Week 16: number analyzed (Participants) | 7
  Week 16 | -0.036 (0.312)
  Week 36: number analyzed (Participants) | 5
  Week 36 | -0.075 (0.244)
  Week 52: number analyzed (Participants) | 4
  Week 52 | 0.031 (0.483)

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: Adverse event (AE): any untoward medical occurrence in a participant who received investigational medicinal product (IMP) without regard to possibility of causal relationship with the treatment. TEAEs: AEs that developed/worsened or became serious during treatment-emergent period (time of first dose administration of study medication up to 28 days after last dose). Serious AE (SAE): any untoward medical occurrence resulted in any of following outcomes: death, life-threatening, required initial/prolonged in-patient hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event.
Time Frame: From first dose administration (i.e., Day 1) of study medication up to 28 days after last dose (i.e., up to 57.5 weeks)
Population: Analysis was performed on safety population which included all participants who received at least 1 dose of belumosudil 200 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil
Number analyzed (Participants) | 10
Participants
  Any TEAEs | 10
  Any TESAEs | 4

ADVERSE EVENTS:
Time Frame: From first dose administration (i.e., Day 1) of study medication up to 28 days after last dose (i.e., up to 57.5 weeks)
Description: Reported AEs and deaths were treatment emergent AEs that developed, worsened, or became serious during treatment emergent period (time from first dose of study drug up to 28 days after the last dose of study drug). Analysis was performed on safety population.
Arm/Group | Belumosudil
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belumosudil (N=10)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belumosudil (N=10)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 1 (1)
Dry Eye (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 2 (2)
Vision Blurred (Eye disorders) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (9)
Oral Pain (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Tooth Discolouration (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (8)
Fatigue (General disorders) | 5 (7)
Pyrexia (General disorders) | 1 (2)
Covid-19 (Infections and infestations) | 2 (2)
Coronavirus Infection (Infections and infestations) | 2 (2)
Gastrointestinal Bacterial Overgrowth (Infections and infestations) | 1 (2)
Helicobacter Gastritis (Infections and infestations) | 1 (1)
Helicobacter Infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (6)
Oral Candidiasis (Infections and infestations) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1)
Rash Pustular (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1)
Urine Analysis Abnormal (Investigations) | 1 (1)
Weight Decreased (Investigations) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (3)
Temporomandibular Joint Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Memory Impairment (Nervous system disorders) | 2 (2)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1)
Abnormal Dreams (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Breast Mass (Reproductive system and breast disorders) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Skin Tightness (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Raynaud's Phenomenon (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Due to slow enrollment and strategic consideration, Sponsor decided to terminate the study and the termination was not driven by any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT04680975/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT04680975/SAP_001.pdf